CLINICAL TRIAL: NCT01446731
Title: Dendritic Cell Vaccination in Combination With Docetaxel for Patients With Cancer Prostate - a Randomized Phase II Study
Brief Title: Dendritic Cell Vaccination and Docetaxel for Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UR1121
Record Dates: First submitted 2011-10-02; First posted 2011-10-05 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-01

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): DC vaccine (mRNA transfected dendritic cell) + Docetaxel
  Interventions: Biological: mRNA transfected dendritic cell; Drug: Docetaxel
- Arm B (Active Comparator): Docetaxel alone
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: mRNA transfected dendritic cell — Autologous monocytes are matured into dendritic cells which are then transfected with mRNA from PSA, PAP, survivin and hTERT.
  5x 10e6 DCs are given as intradermal injections in the groin Day 8 and Day 15 in a 3 week period repeated 4 times and thereafter Day 8 in a 3 week period until progression (no maximum duration).
  Arms: Arm A
Drug: Docetaxel — Docetaxel 75 mg/m2 is given as an intravenous injection Day 1 every three weeks in a maximum of 12 cycles (1 cycle = 3 weeks).
  Other Names: taxotere

SUMMARY:
This is a randomized phase II trial including 40 patients with castration resistant metastatic cancer prostate (CRMPC).

Patients will be randomized between treatment with a dendritic cell vaccine plus docetaxel and docetaxel alone.

The primary objective is to evaluate the vaccine specific immune response and patients will be evaluated with blood tests and DTH reactions during the treatment course.

Secondary objectives are to evaluate clinical response by objective response (RECIST-criteria, 18F-NaF-PET/CT scan), PSA response, pain response and finally we determine time to progression and overall survival.

DETAILED DESCRIPTION:
Treatment in details:

Dendritic cell (DC) vaccination The DC vaccine consists of adherent monocytes collected by leukapheresis. Monocytes are stimulated with GM-CSF and IL-4, and IL-1β, TNFα, IL-6 and PGE2 are used for further maturation.

DCs are transfected with PSA, PAP, survivin and hTERT mRNA. DC vaccines will only be given to patients in ARM A

Docetaxel:

Docetaxel will be given as an i.v. infusion every third week, 75 mg/m2 according to standard treatment. Patients will be pretreated with prednisolon before infusion with Docetaxel. Continuous treatment with prednisolon will not be administered.

Treatment schedule:

The DC vaccination will be administered once a week in two out of three weeks for the first 12 weeks. After 12 weeks the DC vaccination will be given once every three weeks as long as Docetaxel is given. If the disease does not progress but the patient stop treatment with Docetaxel (because of side effects) the vaccine treatment can continue until disease progression.

Evaluation in details:

Immunological evaluation:

Blood tests:

100 ml blood will be drawn from the patient together with the first (baseline), the third and the fourth infusion of Docetaxel, and every third month thereafter.

DTH:

DTH with 3 i.d. injections consisting of media (neg. test), naked DCs and mRNA transfected DCs will be performed at baseline (together with 1st vaccine), together with the 5th vaccine and after three months of treatment (8th vaccine). 48 hours after the DTH at 5th vaccine a biopsy will be taken from the DTH area.

Clinical evaluation:

PSA:

Patients will be evaluated with PSA measurements during the treatment. All patients will receive at least 4 treatments with Docetaxel even if PSA is rising.

18F-NaF ("bone") PET/CT scan: All patients will have a bone-PET/CT scan at baseline. For patients with measurable lesions a PET/CT scan will be performed every three months.

ELIGIBILITY:
Inclusion Criteria:

1. Histological verified CRMPC in progression, defined by

   1. RECIST-criteria and/or
   2. PSA increase to more than baseline in two consecutive measurements
2. Treatment with Docetaxel is indicated
3. Age > 18 years old
4. ECOG performance status ≤2
5. Life expectancy > 3 months
6. Normal organ function

Exclusion Criteria:

1. Other malignant tumors
2. Severe heard or lung disorders
3. Infection with HIV, hepatitis, tuberculosis.
4. Severe allergy or previous anaphylactic reactions
5. Active autoimmune disease
6. Treatment with immunosuppressive drugs (including prednisolon, methotrexate)7. Co-treatment with other experimental treatments, other antineoplastic treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Kongsted, MD, Principal Investigator — CCIT / Department of Oncology, Herlev Hospital
Locations (2):
- Denmark (2):
  - Center for Cancer Immune Therapy, Dept. of Haematology/Oncology, Copenhagen, Herlev
  - Department of Oncology, Herlev Hospital, Herlev

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: DC vaccine + Docetaxel
  mRNA transfected dendritic cell: Autologous monocytes are matured into dendritic cells which are then transfected with mRNA from PSA, PAP, survivin and hTERT.
  5x 10e6 DCs are given as intradermal injections in the groin Day 8 and Day 15 in a 3 week period repeated 4 times and thereafter Day 8 in a 3 week period until progression (no maximum duration).
  Docetaxel: Docetaxel 75 mg/m2 is given as an intravenous injection Day 1 every three weeks in a maximum of 12 cycles (1 cycle = 3 weeks).
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 22 | 21
Completed | 21 | 19
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm A: DC vaccine (mRNA transfected dendritic cell) + Docetaxel
  mRNA transfected dendritic cell: Autologous monocytes are matured into dendritic cells which are then transfected with mRNA from PSA, PAP, survivin and hTERT.
  5x 10e6 DCs are given as intradermal injections in the groin Day 8 and Day 15 in a 3 week period repeated 4 times and thereafter Day 8 in a 3 week period until progression (no maximum duration).
  Docetaxel: Docetaxel 75 mg/m2 is given as an intravenous injection Day 1 every three weeks in a maximum of 12 cycles (1 cycle = 3 weeks).
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 20 | 18 | 38
Age, Continuous [Median (Full Range); unit: years] | 71 [63 to 80] | 70 [60 to 84] | 71 [60 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 21 | 19 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 19 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Immunological Response
Description: The induction of vaccine specific immune responses will be assessed using interferon-gamma ELISPOT assay
Time Frame: 2 years
Population: Biological material for testing was available for 18 patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A
Number analyzed (Participants) | 18
Participants | 9

2. Secondary Outcome: Number of Patients With PSA Response
Description: PSA response will be evaluated by PSA measurements. A 50% decline in PSA is considered to be a response.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 21 | 19
Participants | 11 | 8

3. Secondary Outcome: Number of Patients With Adverse Event Considered Related to the Dendritic Cell Vaccine
Description: Graded according to common terminology criteria for adverse events (CTCAE) version 3.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A
Number analyzed (Participants) | 21
Participants | 2

4. Secondary Outcome: Progression-free Survival
Description: PFS was defined as the time from initiation of docetaxel to clinical, radiographic and/or PSA progression or death. PFS was described using the Kaplan-Meier method.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 21 | 19
months | 5.7 [1.7 to 9.7] | 5.5 [4.8 to 6.2]

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 3/21 | 1/19
Other Adverse Events (participants affected / at risk) | 21/21 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=21) | Arm B (N=19)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Admitted with abdominal pain. Scan showed no ileus. Condition relieved with laxatives.
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=21) | Arm B (N=19)
Allergic reaction (Immune system disorders) | 6 (6) | 2 (2)
Fatigue (General disorders) | 18 (18) | 16 (16)
Weigt loss (General disorders) | 6 (6) | 3 (3)
alopecia (Skin and subcutaneous tissue disorders) | 17 (17) | 18 (18)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Vision impairment (Eye disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 7 (7) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (13) | 14 (14)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 7 (7)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 11 (11) | 14 (14)
Edema limbs (General disorders) | 2 (2) | 4 (4)
Injection site reaction (General disorders) | 2 (2) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
White blood cell decreased (Blood and lymphatic system disorders) | 6 (6) | 3 (3)
Neutrophil count decreased (Blood and lymphatic system disorders) | 6 (6) | 5 (5)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes